CLINICAL TRIAL: NCT04963244
Title: Biomarker of Acute Exacerbation of COPD
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-099
Record Dates: First submitted 2021-06-07; First posted 2021-07-15 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: COPD Exacerbation
Keywords: chronic obstructive pulmonary disease; acute exacerbation; transcriptomic; pathogenesis; biomarkers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AECOPD
- Stable COPD
- Control

INTERVENTIONS:
Other:

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) is the main factor that leads to the deterioration of the disease. Currently, the diagnosis of AECOPD mainly relies on clinical manifestations, and good predictors or biomarkers are lacking. This study aims to explain the gene expression changes related to the disease at the transcriptional level and validate it in multiple levels, reveal specific biomarkers and potential pathogenesis, to provide a research basis for the diagnosis and treatment of AECOPD.

ELIGIBILITY:
For stable COPD:

Inclusion Criteria:

1. Over 40 years old.
2. in line with the diagnostic criteria in GOLD 2018.
3. with the ability to sign informed consent.
4. can be followed up according to the study protocol.

Exclusion Criteria:

1. with other pulmonary diseases (such as lung cancer, sarcoidosis, tuberculosis, pulmonary fibrosis, cystic fibrosis) and severe α1-antitrypsin deficiency.
2. with other inflammatory diseases (such as rheumatoid arthritis and inflammatory bowel disease, etc.).
3. a history of pulmonary surgery, or a diagnosis of malignant tumor recently.
4. a history of blood transfusion in 4 weeks.
5. participating in a double-blind drug clinical trial.
6. unable to walk.
7. using oral or intravenous steroid therapy.
8. with acute exacerbation in 4 weeks.

For AECOPD:

Inclusion Criteria:

Patients who were over 40 years old were eligible for inclusion if they had a diagnosis of COPD in their primary care clinical record and were presenting with an acute exacerbation of respiratory symptoms.

Exclusion Criteria:

1. Other specific diseases that may account for sudden changes in respiratory symptoms should be excluded by clinical or laboratory tests.
2. The remaining exclusion criteria were consistent with the above five criteria in stable COPD.

The control group:

Inclusion Criteria:

Healthy people over 40 years old.

Exclusion Criteria:

with chronic airway diseases and other lung diseases, and heart, kidney, liver, and other important organ diseases.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stable COPD and AECOPD and healthy controls were recruited from the Second Affiliated Hospital of Zhejiang University School of Medicine and Yuhang District of the Second Affiliated Hospital of Zhejiang University, Hangzhou, China.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Differentially expressed genes of 13 participants as assessed by RNA sequencing | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China